CLINICAL TRIAL: NCT02481401
Title: Family-based Approach in a Minority Community Integrating Systems-Biology for Promotion of Health
Brief Title: Family-based Approach to Promotion of Health - FAMILIA (Project 2)
Acronym: FAMILIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 14-0256 Project 2
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Promoting Cardiovascular Health in Adults; Lifestyle Intervention; Atherosclerosis
Keywords: cardiovascular health; behavior change; community-based; family-based; prevention
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Will not receive any structured program except for the health promotion education program that the children will receive for 4 months. Complementary to the Si! Program. This is essentially healthy habits related information and activities to be performed with their kids through family newsletters. All participants (including controls) have access to the study website for health related information.
- Intensive Individual Intervention Program (Experimental): A combination of one-on-one personalized lifestyle counseling (8 months with 4 complimentary sessions for a total of 12 months) and a wearable physical activity monitor such as the Garmin Vivofit.
  Interventions: Behavioral: Intensive Individual Intervention Program
- Peer-To-Peer Program Intervention (Active Comparator): Monthly meetings for 60-90 minutes in groups of about up to 20 supporting each other in self-control of CV risk factors, for a total of 12 months.
  Interventions: Behavioral: Peer-To-Peer Program Intervention

INTERVENTIONS:
Behavioral: Intensive Individual Intervention Program
  Arms: Intensive Individual Intervention Program
Behavioral: Peer-To-Peer Program Intervention
  Arms: Peer-To-Peer Program Intervention

SUMMARY:
Two Intensive Life Style Intervention Programs in Related Caregivers of Preschool Children

Substantial strides have been made in the treatment of acute cardiovascular conditions, such as myocardial infarction and stroke, however, the global burden of cardiovascular disease (CVD) continues to rise at an alarming rate. Furthermore, despite the abundant data demonstrating a greater burden of CVD in racial/ethnic minorities, and many specific interventions aimed at changing risk factor patterns or behaviors in racial/ethnic minorities, health disparities persist. In the present study, the investigators seek to evaluate the impact of a multifaceted and comprehensive lifestyle intervention coupled with atherosclerosis imaging on reducing cardiovascular risk among minority adults living in Harlem, New York. The investigators believe that holistic, multi-dimensional individual and peer-to-peer intensive lifestyle interventions involving parents/caregivers of preschool children will be effective in producing favorable change in their behaviors, which will be sustained over time. The primary hypothesis of the study is that aggressive lifestyle interventions will be more effective in improving healthy behaviors and biological correlates in at-risk adult parents and/or caregivers of preschool children in Harlem, NY. In aim 1, as an initial pilot study, the investigators will identify the contextual factors, facilitators and barriers that may impact the implementation of a lifestyle intervention program for adults in Harlem, using qualitative research methods. In aim 2, the investigators will determine the impact of two intensive lifestyle interventions on promoting and improving healthy behaviors and biological parameters to lower cardiovascular risk, the impact of the knowledge of presence of atherosclerosis on health behaviors and the impact of these lifestyle interventions on atherosclerosis among approximately 600 asymptomatic at-risk adults. Finally, in aim 3, the investigators will evaluate the sustainability of the impact of the two intensive lifestyle interventions on healthy behaviors and biological parameters approximately 12 months after the intervention program ends.

DETAILED DESCRIPTION:
Aim 1 - Pilot: To identify the contextual factors, facilitators and barriers that may impact the implementation of a lifestyle intervention program for adults in Harlem, using qualitative research methods: 1) focus group discussions among a representative cohort of adults; 2) focus group discussions among community leaders; and 3) Pilot studies of feasibility of interventions in the representative cohort of adults.

Subsidiary Aim 1.1: To use identified facilitators and barriers to develop a contextually and culturally appropriate model for an adult lifestyle intervention program.

Subsidiary Aim 1.2: To implement a pilot intervention of the contextually and culturally adapted program among a sample of parents/caregivers of children in preschools in Harlem.

The investigators will assess for acceptability and feasibility, and make any necessary modifications prior to the implementation of the cluster-randomized trial. This aim will be carried out at 2 preschools in Harlem, NY by including the parents and caregivers of pre-school children. The final intervention program that results from this intervention-mapping program will be piloted in parent groups of 8-10.

Aim 2 - Randomization: To determine (i) the impact of two intensive lifestyle interventions on promoting and improving healthy behaviors (increased physical activity, smoking cessation etc.) and biological parameters (lipids, sugar) to lower cardiovascular risk, (ii) the impact of the presence of atherosclerosis on health behaviors and (iii) the impact of the lifestyle interventions on atherosclerosis among approximately 600 asymptomatic at-risk adults.

Hypothesis: Adults receiving the lifestyle intervention programs will demonstrate a greater improvement in healthy behaviors and biological parameters compared to controls.

Hypothesis: Knowledge of presence of atherosclerosis as defined by three-dimensional vascular ultrasound will lead to greater improvement in healthy behaviors.

Hypothesis: Adults receiving the lifestyle intervention programs will demonstrate a lesser progression or regression of three-dimensional vascular ultrasound quantified atherosclerosis compared to controls.

For this aim, the investigators will recruit parents and caregivers of pre-school children from up to twenty schools in Harlem, NY and perform a 3:2 (3 intervention, 2 control) cluster randomization of the schools. Those schools in the "intensive intervention" group will be randomly assigned to one of two interventions- an Intensive Individual Intervention Program" (IIIP) developed through the intervention mapping program described in aim 1 or 'Peer-To-Peer Program - Intervention" (PPPI), refined during that same pilot phase. The primary outcome will be a composite score consisting of a 0-3 scale for behaviors/outcomes related to Blood pressure, Exercise, Weight, Alimentation (diet) and Tobacco (smoking) [Fuster-BEWAT score]. Primary assessments will be performed at baseline, at the end of the intervention (approximately 12 months, peak effect), and at approximately 24 months (sustainability). The 12 month assessment will be used to calculate the between group difference for the change in the Fuster-BEWAT score and will be the primary outcome measure for the adults. To evaluate the sustainability of the impact of the two intensive lifestyle interventions on healthy behaviors and biological parameters 12 months after the intervention program ends. For the assessment of secondary outcome measures, participants will undergo point of care testing for a lipid panel and blood sugar assessment, and a three-dimensional vascular ultrasound (carotid, ileo-femoral) to assess for presence and extent of atherosclerosis at baseline and after the intervention period.

Blood will be collected from all adults who provide consent at enrollment and at the end of the intervention period. Blood from adults will be used to isolate DNA and plasma. In addition, by in vitro culture of blood-derived mononuclear cells, we will derive macrophages, which will then be driven to become foam cells. RNA will be isolated from pre- and post-intervention blood samples. Genomic data obtained from adult blood samples will be integrated with data obtained from saliva in children to identify network models and predictors of primary prevention outcomes. Also, RNA data will be integrated to identify the genetic, genomic and molecular signature of favorable vs. poor responders to lifestyle intervention; and to identify novel therapeutic and diagnostic targets in network models of early atherothrombotic disease.

Aim 3 - Sustainability: To evaluate the sustainability of the impact of the two intensive lifestyle interventions on healthy behaviors and biological parameters approximately 12 months after the intervention program ends.

Hypothesis: Adult caregivers receiving the intensive lifestyle approaches program, will maintain sustainability with an advantage of the two "Intensive Interventional groups" over the control "Traditional Health Education" group. All participants will be followed for approximately 12 months after the end of the intervention period and reassess their Fuster-BEWAT Score.

ELIGIBILITY:
Inclusion Criteria:

Parents and caretakers of children attending 15 preschools that will be comparable in characteristics related to socio-economic level and ethnicity.

* The schools must be located in Harlem, NY.
* The schools must be public.
* The schools must have children 3, 4 and 5 years of age.
* The schools must provide meals for the children.
* The schools must make available use of their applicable program operation space.

Adult parents and/or caregivers of children enrolled in the FAMILIA children's study will be approached for participation in this study.

Exclusion Criteria:

* Participation in any other major structured health intervention program similar to the FAMILIA Program during the evaluation of the program.
* Inability to carry out all activities proposed by the FAMILIA Program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2015-11; Primary Completion 2018-06 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Fuster-BEWAT Score | baseline and 12 months
  BEWAT stands for Blood pressure, Exercise, Weight, Alimentation (diet) and Tobacco (smoking). Change in Fuster-BEWAT score at 12 months as compared to baseline. The overall BEWAT scale ranges from 0 (poor health) to 15 (ideal cardiovascular health). Higher score indicates healthier outcomes.

SECONDARY OUTCOMES:
Change in Fuster-BEWAT Score | Baseline and 24 months
  BEWAT stands for Blood pressure, Exercise, Weight, Alimentation (diet) and Tobacco (smoking). The overall BEWAT scale ranges from 0 (poor health) to 15 (ideal cardiovascular health). Higher score indicates healthier outcomes.
Change in individual domains assimilated in the composite Fuster-BEWAT Score | Baseline and 12 months
  BEWAT stands for Blood pressure, Exercise, Weight, Alimentation (diet) and Tobacco (smoking). The individual domain score for physical activity (range 0-3), fruit and vegetable consumption (range 0-3), body-mass index (range BMI) (0-3), smoking habits (range 0-3), and blood pressure (range 0-3). Higher score indicates healthier outcomes.
Change in individual domains assimilated in the composite Fuster-BEWAT Score | Baseline and 24 months
  BEWAT stands for Blood pressure, Exercise, Weight, Alimentation (diet) and Tobacco (smoking). The individual domain score for physical activity (range 0-3), fruit and vegetable consumption (range 0-3), body-mass index (range BMI) (0-3), smoking habits (range 0-3), and blood pressure (range 0-3). Higher score indicates healthier outcomes.
Change in Blood Pressure | baseline and 12 months
  Change in blood pressure at 12 months as compared to baseline
Change in Blood Pressure | baseline and 24 months
  Change in blood pressure at 24 months as compared to baseline
Change in IPAQ | baseline and 12 months
  International Physical Activity Questionnaire (IPAQ). Change in IPAQ at 12 months as compared to baseline. It is measured as a continuous variable based on length of time. and expressed as MET-min per week: MET level x minutes of activity x events per week.
Change in IPAQ | baseline and 24 months
  Change in IPAQ scale at 24 months as compared to baseline. IPAQ stands for International Physical Activity Questionnaire. It is measured as a continuous variable based on length of time. and expressed as MET-min per week: MET level x minutes of activity x events per week.
Change in plaque volume | baseline and 12 months
  Change in plaque volume at 12 months as compared to baseline
Change in blood lipid profile | baseline and 12 months
  Change in blood lipid profile at 12 as compared to baseline.
Change in blood lipid profile | baseline and 24 months
  Change in blood lipid profile at 24 months as compared to baseline.
Change in blood glucose | baseline and 12 months
  Change in blood glucose at 12 months as compared to baseline.
Change in blood glucose | baseline and 24 months
  Change in blood glucose at 24 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Study Director — Icahn School of Medicine at Mount Sinai; Zahi Fayad, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - Lutheran Social Services, Site 14, New York, New York
  - West Harlem Community Organization, Inc., New York, New York
  - East Harlem Community Organization, Inc., Site 2, New York, New York
  - East Harlem Council for Human Services, Inc., Site 1, New York, New York
  - Union Settlement Carver Childcare Center, New York, New York
  - Union Settlement Head Start at Franklin Plaza, New York, New York
  - Union Settlement Johnson, New York, New York
  - Union Settlement Leggett Memorial, New York, New York
  - Union Settlement Washington, New York, New York
  - Addie Mae Collins Head Start, Site 1, New York, New York
  - Addie Mae Collins Head Start, Site 2, New York, New York
  - Addie Mae Collins Head Start, Site 3, New York, New York
  - Association to Benefit Children Graham School, New York, New York
  - Lutheran Social Services, Site 11, New York, New York
  - Lutheran Social Services, Site 12, New York, New York

REFERENCES:
- [Background] Vedanthan R, Bansilal S, Soto AV, Kovacic JC, Latina J, Jaslow R, Santana M, Gorga E, Kasarskis A, Hajjar R, Schadt EE, Bjorkegren JL, Fayad ZA, Fuster V. Family-Based Approaches to Cardiovascular Health Promotion. J Am Coll Cardiol. 2016 Apr 12;67(14):1725-37. doi: 10.1016/j.jacc.2016.01.036. PMID 27056780
- [Background] Bansilal S, Vedanthan R, Kovacic JC, Soto AV, Latina J, Bjorkegren JLM, Jaslow R, Santana M, Sartori S, Giannarelli C, Mani V, Hajjar R, Schadt E, Kasarskis A, Fayad ZA, Fuster V. Rationale and Design of Family-Based Approach in a Minority Community Integrating Systems-Biology for Promotion of Health (FAMILIA). Am Heart J. 2017 May;187:170-181. doi: 10.1016/j.ahj.2017.02.020. Epub 2017 Feb 22. PMID 28454800
- [Derived] Iglesies-Grau J, Fernandez-Jimenez R, Diaz-Munoz R, Jaslow R, de Cos-Gandoy A, Santos-Beneit G, Hill CA, Turco A, Kadian-Dodov D, Kovacic JC, Fayad ZA, Fuster V. Subclinical Atherosclerosis in Young, Socioeconomically Vulnerable Hispanic and Non-Hispanic Black Adults. J Am Coll Cardiol. 2022 Jul 19;80(3):219-229. doi: 10.1016/j.jacc.2022.04.054. PMID 35835495